CLINICAL TRIAL: NCT02415972
Title: Dynamic Contrast-enhanced Ultrasound Imaging for Cerebral Perfusion Measurement in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 179/12
Record Dates: First submitted 2015-03-27; First posted 2015-04-14 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Acute Ischemic Stroke
Keywords: ultrasound imaging; acute ischemic stroke; cerebral perfusion measurement in acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Patients with Stroke
  Interventions: Other: Ultrasound perfusion imaging

INTERVENTIONS:
Other: Ultrasound perfusion imaging — Dynamic perfusion imaging of brain parenchyma with modern ultrasound is possible with the use of ultrasound contrast media that serve as echo signal amplifier.

SUMMARY:
Stroke, a personal, familial, and social disaster, is the first cause of acquired disability, the second cause of dementia, and the third cause of death worldwide. Its associated socio-economic costs are astronomic. The burden of stroke is likely to increase, given the aging of the population and the growing incidence of many vascular risk factors. Therefore, apart from further development of stroke prevention and treatment strategies, rational and effective tools for diagnosis, monitoring, and follow-up for stroke patients have potential high long-term clinical and economic consequences.

For neuroradiological work-up, computed tomography (CT) or magnetic resonance imaging (MRI) are used as gold standard techniques to detect presence or absence, effective state, and extent of stroke. However, these techniques achieve simply a baseline study of ischemia occurred and can deliver only a snapshot of brain parenchyma and vessels. Furthermore, their rapid and actual availability, especially in primary hospitals, and their dynamic capabilities and predictive values for further infarction are poor with critically ill patients have to be repeatedly transferred to the scanning unit for each measurement. Whereas CT examination is associated with x-ray radiation and may miss early detection of stroke, MRI is associated with higher costs and not generally routinely and around-the clock available in all the hospitals. Therefore, a simple, fast, repeatable, non-hazardous, and non-invasive dynamic bedside tool for the detection of acute brain tissue hypoperfusion and monitoring for potential further infarction or efficacy of thrombolysis either by systemic intravenous thrombolytic therapy with recombinant tissue plasminogen activator (rt-PA) or by selective intraarterial fibrinolysis and mechanical recanalization, both combined with or without bridging after acute ischemic stroke, is strongly needed.

A promising alternative method of diagnosing stroke represents contrast-enhanced ultrasound perfusion imaging (UPI). What makes UPI so valuable is the advantage of repeatedly and non-invasively detecting brain tissue at risk for infarction by dynamic direct brain tissue perfusion assessment and not by surrogate parameters, like blood flow velocity or vessel diameter. Because of the possibility to screen and repeatedly measure the state of perfusion, the chances increase to diagnose and monitor ischemic stroke and to define the appropriate window for treatment. The perfusion analysis would also allow determination of treatment results and guidance of rapid and adequate further therapy.

Therefore, the present pilot study in 40 patients is initiated. The objectives of this observational diagnostic cohort trial are to evaluate feasibility and practicability of repeated bedside assessments by contrast enhanced UPI in acute ischemic stroke patients and to assess whether UPI can detect alterations in brain tissue perfusion before and after recanalising therapy of strokes. Assessment of cerebral perfusion by CT or MRI serves as reference and its results are compared to UPI data.

DETAILED DESCRIPTION:
Background

Stroke is a personal, familial and social disaster. Apart from development of stroke prevention and treatment strategies, the mainstay of stroke research remains new-product development and improvement of current imaging tools for diagnosis, monitoring and follow-up of stroke patients. For initial neuroradiological work-up, usually computed tomography (CT) or magnetic resonance imaging (MRI) are used to detect presence or absence, effective state and extent of stroke. However, their rapid and actual availability, especially in primary hospitals, and their dynamic capabilities and predictive values for further infarction are poor. Currently cerebral CT-perfusion (CTP) imaging can be regarded as the gold standard for assessing tissue hypoperfusion in this setting. It employs, however, both contrast agent and X-ray exposition and patients have to be repeatedly transferred to the scanning unit for each measurement. Therefore, a fast, simple, repeatable, non-hazardous and non-invasive dynamic bedside tool for the detection of acute brain tissue hypoperfusion and monitoring for potential further infarction or efficacy of thrombolysis after ischemic stroke is strongly needed.

Socioeconomic importance of stroke Stroke is the first cause of acquired disability, the second cause of dementia and the third cause of death worldwide, and its associated socio-economic costs are astronomic. The burden of stroke is likely to increase, given the aging of the population and the growing incidence of many vascular risk factors. Therefore, rational and effective diagnostic and therapeutic management in stroke patients has potential high long-term clinical and economic consequences.

Current standard therapy after acute ischemic stroke According to the cause of stroke and apart from medical treatment and surgical options in selected cases, the mainstay of therapeutic management of acute ischemic stroke itself usually remain systemic intravenous thrombolytic therapy with recombinant tissue plasminogen activator (rt-PA) or selective intraarterial fibrinolysis and mechanical recanalization, both with or without bridging (combined intravenous and intraarterial thrombolysis). In this regard, reperfusion therapy is the only proven treatment for acute ischemic stroke.

Current problems in diagnosis and monitoring of stroke patients At present, CT and MRI are usually applied for diagnosis and follow-up of stroke. However, both CT and MRI achieve simply a baseline study of ischemia occurred and can deliver only a snapshot of brain parenchyma and vessels. Furthermore, whereas CT examination is associated with x-ray radiation and may miss early detection of stroke, MRI is associated with higher costs and is not generally routinely and around-the clock available in all the hospitals. Both imaging methods require transportation and intensive care of the often critically ill patients to the scanning unit for each measurement.

There is unanimous agreement about the need for a bedside assessment of the status of tissue perfusion. Invasive cerebral angiography is indicated in cases of further evaluation of stroke causes and intended endovascular therapy.

Potential of ultrasound perfusion imaging (UPI) What makes contrast enhanced UPI so valuable is the possibility to repeatedly and non-invasively detect brain tissue at risk for infarction by direct brain tissue perfusion assessment and not by surrogate parameters, like blood flow velocity or vessel diameter. Because of the possibility to screen and repeatedly measure the state of perfusion, the chances increase to diagnose and monitor ischemic stroke and to define the appropriate window for treatment. The perfusion analysis would also allow determination of treatment results and guidance of rapid and adequate further therapy.

Objective

The objective of the present study is to assess whether cerebral hypoperfusion can be detected by ultrasound perfusion imaging (UPI) before and after treatment of acute ischemic stroke.

Methods

Patients with acute middle cerebral artery (MCA) territory ischemic stroke are evaluated for potential thrombolysis/thrombectomy according to the Bernese neurologic stroke algorithm. An experienced neurosonographer performs contrast-enhanced ultrasound perfusion imaging (UPI) after prospective study enrollment and specific stroke CT/MRI with perfusion measurement. Clinical status is documented by use of the NIHSS on admission /first day after the intervention. UPI and CT/MRI perfusion data is analyzed. Two different quantification algorithms, standard versus patient-adjusted, are used. Data is analyzed by descriptive statistics using the mean, median and standard deviation of the ROIs. Sensitivity and specificity analyses are calculated using Pearson's chi-square test. Receiver-operator characteristic curves are calculated for UPI/perfusion MRI/CT parameters. Pearson correlation is used to evaluate correlations between absolute values of UPI and MRI TTP data.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an indication for iv thrombolysis or endovascular treatment according to the current stroke guidelines of the University Hospital Bern
* Age ≥18
* Written informed consent by patient or next of kin
* Signed consent of independent physician

Exclusion Criteria

* Positive pregnancy test and breast feeding
* Acute coronary syndromes, severe ischemic heart disease (requiring revascularization), severe aortic and mitral valve disease, severe congestive heart failure (NYHA >III/IV)
* Severe pulmonary or renal dysfunction
* Known allergy or adverse reaction to contrast material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial population comprises of patients with acute ischemic stroke treated at the University Hospital Bern.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with detection of cerebral hypoperfusion before and after thrombolytic treatment and correlation to established diagnostic gold standard CT- or MRI-perfusion studies by measurement of time to peak values | 1 day after intervention

SECONDARY OUTCOMES:
Number of Patients with Adverse Events as a Measure of Safety and Tolerability and detection of early clinical outcome by NIHSS | 1 day after intervention
Quantitative analysis of metric parameters of UPI | 1 day after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Beck, Prof. Dr. med., Principal Investigator — Department of Neurosurgery, Bern University Hospital Bern
Locations (1):
- Department of Neurosurgery, Bern University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Beck J, Raabe A, Lanfermann H, Seifert V, Weidauer S. Tissue at risk concept for endovascular treatment of severe vasospasm after aneurysmal subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1779-81. doi: 10.1136/jnnp.2004.036921. PMID 15548506
- [Background] Beck J, Raabe A, Lanfermann H, Berkefeld J, De Rochemont Rdu M, Zanella F, Seifert V, Weidauer S. Effects of balloon angioplasty on perfusion- and diffusion-weighted magnetic resonance imaging results and outcome in patients with cerebral vasospasm. J Neurosurg. 2006 Aug;105(2):220-7. doi: 10.3171/jns.2006.105.2.220. PMID 17219826
- [Background] Beck J, Raabe A, Lanfermann H, Seifert V, Weidauer S. Perfusion-weighted magnetic resonance imaging in patients with vasospasm: a useful new tool in the management of patients with subarachnoid hemorrhage. Neurosurgery. 2006 Mar;58(3):E590; author reply E590. doi: 10.1227/01.NEU.0000207963.98939.7B. No abstract available. PMID 16528172
- [Background] Eyding J, Krogias C, Schollhammer M, Eyding D, Wilkening W, Meves S, Schroder A, Przuntek H, Postert T. Contrast-enhanced ultrasonic parametric perfusion imaging detects dysfunctional tissue at risk in acute MCA stroke. J Cereb Blood Flow Metab. 2006 Apr;26(4):576-82. doi: 10.1038/sj.jcbfm.9600216. PMID 16121127
- [Background] Seidel G, Meyer-Wiethe K, Berdien G, Hollstein D, Toth D, Aach T. Ultrasound perfusion imaging in acute middle cerebral artery infarction predicts outcome. Stroke. 2004 May;35(5):1107-11. doi: 10.1161/01.STR.0000124125.19773.40. Epub 2004 Mar 18. PMID 15031454
- [Background] Wiesmann M, Meyer K, Albers T, Seidel G. Parametric perfusion imaging with contrast-enhanced ultrasound in acute ischemic stroke. Stroke. 2004 Feb;35(2):508-13. doi: 10.1161/01.STR.0000114877.58809.3D. Epub 2004 Jan 22. PMID 14739406
- [Background] Kern R, Diels A, Pettenpohl J, Kablau M, Brade J, Hennerici MG, Meairs S. Real-time ultrasound brain perfusion imaging with analysis of microbubble replenishment in acute MCA stroke. J Cereb Blood Flow Metab. 2011 Aug;31(8):1716-24. doi: 10.1038/jcbfm.2011.14. Epub 2011 Mar 2. PMID 21364598
- [Background] Eyding J, Krogias C, Meves S, Przuntek H, Postert T. Quantitative ultrasonographic evaluation of cerebral perfusion in acute stroke is possible. Stroke. 2004 Nov;35(11):2432-3; author reply 2433. doi: 10.1161/01.STR.0000143731.48504.7d. Epub 2004 Sep 16. No abstract available. PMID 15375306
- [Background] Engelhardt M, Hansen C, Eyding J, Wilkening W, Brenke C, Krogias C, Scholz M, Harders A, Ermert H, Schmieder K. Feasibility of contrast-enhanced sonography during resection of cerebral tumours: initial results of a prospective study. Ultrasound Med Biol. 2007 Apr;33(4):571-5. doi: 10.1016/j.ultrasmedbio.2006.10.007. PMID 17337111
- [Background] Kopp R, Zurn W, Weidenhagen R, Meimarakis G, Clevert DA. First experience using intraoperative contrast-enhanced ultrasound during endovascular aneurysm repair for infrarenal aortic aneurysms. J Vasc Surg. 2010 May;51(5):1103-10. doi: 10.1016/j.jvs.2009.12.050. PMID 20420978